CLINICAL TRIAL: NCT04936685
Title: A Phase IIIb, Open-label, Multi-center Study to Evaluate the Immunogenicity and Safety of a Booster Dose and Describe the Immune Persistence of MenACYW Conjugate Vaccine With 5- and/or 10-year Booster Doses in Children and Adolescents Who Had Been Primed With MenACYW Conjugate Vaccine as Toddlers.
Brief Title: Study on an Investigational Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) Administered as a 5- and/or 10-year Booster Doses in Children and Adolescents Vaccinated 5 or 10 Years Earlier as Toddlers
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEQ00073; U1111-1255-4941 (Registry Identifier: ICTRP); 2021-000104-38 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Participants will receive a first booster dose of MenACYW conjugate vaccine at Day 1 and a second booster dose at year 5 of study MEQ00073
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine
- Group 2 (Experimental): Participants will receive a single booster dose of MenACYW conjugate vaccine at year 5 of study MEQ00073
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, W, and Y) Tetanus Toxoid Conjugate Vaccine — Liquid solution for injection Intramuscular
  Other Names: MenACYW conjugate vaccine MenQuadfi®

SUMMARY:
The purpose of the MEQ00073 study is to assess the immunogenicity and safety of a booster dose in children who had been vaccinated with MenACYW conjugate vaccine approximately 5 years earlier as toddlers as part of the MET51 study, and to describe the persistence of a priming dose in children and adolescents who had been vaccinated with MenACYW conjugate vaccine approximately 5 years or 10 years earlier as toddlers as part of the MET51 study, the immunogenicity and safety of a booster dose in adolescents who had been primed with MenACYW conjugate vaccine as toddlers as part of the MET51 study, and the immunogenicity and safety of a second booster dose in adolescents approximately 5 years after a first booster dose as children approximately 5 years after the priming dose as toddlers.

DETAILED DESCRIPTION:
The duration of each participant's participation will be approximately 5.5 years

ELIGIBILITY:
Inclusion Criteria:

* Received MenACYW vaccine in MET51 study (Groups 1 and 3) and completed the study (attended Visit 2)
* Participant and parent/ legally acceptable representative (LAR) are able to attend all scheduled visits and to comply with all trial procedures
* Covered by health insurance, if required by local regulations

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal infection during the trial (specifically but not limited to participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease)
* Personal history of Guillain-Barré syndrome (GBS)
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid containing vaccine
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Verbal report by parent or LAR of thrombocytopenia or suspected thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (ie, mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, W, or Y) with the exception of licensed MenC vaccination received during infancy (MET51 Group 3), of the single dose of meningococcal vaccine administered as part of study MET51 (Group 1 and 3) and of Meningococcal B vaccine
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial vaccination except for influenza vaccination, which may be received at least 2 weeks before or after study vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2027-12-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (26):
- Finland (9):
  - Investigational Site Number : 2460009, Espoo
  - Investigational Site Number : 2460001, Helsinki
  - Investigational Site Number : 2460006, Helsinki
  - Investigational Site Number : 2460002, Jarvenpaa
  - Investigational Site Number : 2460004, Kokkola
  - Investigational Site Number : 2460007, Oulu
  - Investigational Site Number : 2460003, Pori
  - Investigational Site Number : 2460008, Tampere
  - Investigational Site Number : 2460010, Turku
- Germany (9):
  - Investigational Site Number : 2760011, Bönnigheim
  - Investigational Site Number : 2760001, Bramsche
  - Investigational Site Number : 2760007, Bretten
  - Investigational Site Number : 2760004, Erfurt
  - Investigational Site Number : 2760015, Hamburg
  - Investigational Site Number : 2760002, Mönchengladbach
  - Investigational Site Number : 2760008, Mönchengladbach
  - Investigational Site Number : 2760006, Schönau
  - Investigational Site Number : 2760003, Tauberbischofsheim
- Hungary (4):
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480001, Budapest
  - Investigational Site Number : 3480005, Miskolc
  - Investigational Site Number : 3480006, Székesfehérvár
- Spain (4):
  - Investigational Site Number : 7240006, Santiago de Compostela, Galicia [Galicia]
  - Investigational Site Number : 7240001, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240003, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Martinon-Torres F, Simko R, Ebert R, Ramet M, Zocchetti C, Syrkina O, Bchir S, Bertrand-Gerentes I. Five-Year Immune Persistence of a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW-TT) and Immunogenicity and Safety of a Booster Dose in Children. Infect Dis Ther. 2025 May;14(5):991-1010. doi: 10.1007/s40121-025-01121-6. Epub 2025 Apr 1. PMID 40169489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 centers in 4 countries from 23 August 2022 to 06 February 2023.
Pre-assignment Details: A total of 209 participants were enrolled in this study. Results has been reported as per the primary completion date of 09 March 2023. Final analysis results will be reported at a later date.
Groups:
- MenACYW: Group 1: Participants received a first intramuscular (IM) booster dose of 0.5 milliliter (mL) of Meningococcal polysaccharide (Serogroups A, C, Y and W) (MenACYW conjugate vaccine) at Day 1 (visit 1, at child age approximately 5 years post priming dose as toddlers in study MET51) and will receive a second booster dose at Year 5 of the study (visit 3, at adolescent age approximately 5 years post booster dose as children in this study).
- MenACYW: Group 2: Participants will receive a single IM booster dose of 0.5 mL of MenACYW conjugate vaccine at Year 5 (visit 2) of the study (approximately 10 years post priming dose as toddlers in study MET51).
Period: Overall Study
Arm/Group | MenACYW: Group 1 | MenACYW: Group 2
Started | 93 | 116
Completed | 92 | 116
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants with data in Case report form (CRF) consisted of all study participants with CRF, i.e with data in the clinical database.
Groups:
- MenACYW: Group 1: Participants had a blood sample before receiving a first IM booster dose of 0.5 mL of MenACYW conjugate vaccine at Day 1 (visit 1, at child age approximately 5 years post priming dose as toddlers in study MET51).
- MenACYW: Group 2: Participants had a blood sample at Day 1 (Visit 1, at child age approximately 5 years post priming dose as toddlers in study MET51).
- Total: Total of all reporting groups
Arm/Group | MenACYW: Group 1 | MenACYW: Group 2 | Total
Number analyzed (Participants) | 93 | 116 | 209
Age, Continuous [Mean (Standard Deviation); unit: year] | 6.28 (0.578) | 6.26 (0.440) | 6.27 (0.505)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 60 | 95
  Male | 58 | 56 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 93 | 113 | 206
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Group 1: Percentage of Participants With Sufficiency of Serum Bactericidal Assay Using Human Complement (hSBA) Vaccine Seroresponse at 30 Days Post Booster Dose
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. hSBA vaccine seroresponse for serogroups A, C, W, and Y is defined as: percentage of participants with a pre-vaccination titer < 1:8, who had achieved a post-vaccination titer >= 1:16 or participants with a pre-vaccination titer >= 1:8, who had achieved a post-vaccination titer at least 4-fold greater than the pre-vaccination titer. The seroresponse sufficiency was demonstrated if the lower limit of 1-sided 97.5% confidence interval (CI) is > 75%.
Time Frame: Baseline (Day 1) and 30 days after the MenACYW conjugate vaccine 5-year booster dose
Population: The Per-Protocol Analysis Sets 1 (PPAS1) is a subset of the Full analysis set (FAS). The FAS consisted of participants who had received the study vaccine and had a valid post-vaccination serology result 5-years after priming vaccination at visit 1. Participants data whose titers meet the hSBA vaccine seroresponse criteria have been reported.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- MenACYW: Group 1: Participants received a first IM booster dose of 0.5 mL of MenACYW conjugate vaccine at Day 1 (visit 1, at child age approximately 5 years post priming dose as toddlers in study MET51).
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Serogroup A: number analyzed (Participants) | 82
  Serogroup A | 93.2 [85.7 to NA] — Seroresponse sufficiency was demonstrated if the lower limit of 1-sided 97.5% CI was > 75%. Therefore, only 1-sided CI was determined.
  Serogroup C: number analyzed (Participants) | 86
  Serogroup C | 97.7 [92.0 to NA] — Seroresponse sufficiency was demonstrated if the lower limit of 1-sided 97.5% CI was > 75%. Therefore, only 1-sided CI was determined.
  Serogroup W: number analyzed (Participants) | 87
  Serogroup W | 98.9 [93.8 to NA] — Seroresponse sufficiency was demonstrated if the lower limit of 1-sided 97.5% CI was > 75%. Therefore, only 1-sided CI was determined.
  Serogroup Y: number analyzed (Participants) | 87
  Serogroup Y | 98.9 [93.8 to NA] — Seroresponse sufficiency was demonstrated if the lower limit of 1-sided 97.5% CI was > 75%. Therefore, only 1-sided CI was determined.

2. Secondary Outcome: Antibody Persistence of Meningococcal (Groups 1 and 2): Percentage of Participants Achieving Titer (Seroprotection) >=1:8 hSBA and Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Titer >=1:8 Approximately 5 Years After the Primary Vaccination
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA and the rSBA and the results were expressed as vaccine seroprotection. Seroprotection rate is defined as percentage of participants with hSBA titer and rSBA titer >=1.8 who received MenACYW conjugate vaccine 5 years earlier. Antibody persistence of meningococcal serogroups A, C, W, and Y in children at 5 years (Groups 1 and 2).
Time Frame: At Day 1 (approximately 5 year after the administration of a priming dose as toddlers in study MET51)
Population: The FAS3 consisted of participants who had a valid baseline serology results (hSBA or rSBA accordingly). Only data from the participants analyzed were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1 | MenACYW: Group 2
Number analyzed (Participants) | 92 | 116
percentage of participants
  hSBA titer >=1.8, Serogroup A: number analyzed (Participants) | 72 | 86
  hSBA titer >=1.8, Serogroup A | 78.3 [68.4 to 86.2] | 74.1 [65.2 to 81.8]
  hSBA titer >=1.8, Serogroup C: number analyzed (Participants) | 77 | 100
  hSBA titer >=1.8, Serogroup C | 83.7 [74.5 to 90.6] | 86.2 [78.6 to 91.9]
  hSBA titer >=1.8, Serogroup W: number analyzed (Participants) | 78 | 98
  hSBA titer >=1.8, Serogroup W | 84.8 [75.8 to 91.4] | 84.5 [76.6 to 90.5]
  hSBA titer >=1.8, Serogroup Y: number analyzed (Participants) | 66 | 77
  hSBA titer >=1.8, Serogroup Y | 71.7 [61.4 to 80.6] | 66.4 [57.0 to 74.9]
  rSBA titer >=1.8, Serogroup A: number analyzed (Participants) | 66 | 71
  rSBA titer >=1.8, Serogroup A | 71.7 [61.4 to 80.6] | 61.7 [52.2 to 70.6]
  rSBA titer >=1.8, Serogroup C: number analyzed (Participants) | 55 | 68
  rSBA titer >=1.8, Serogroup C | 59.8 [49.0 to 69.9] | 58.6 [49.1 to 67.7]
  rSBA titer >=1.8, Serogroup W: number analyzed (Participants) | 53 | 65
  rSBA titer >=1.8, Serogroup W | 57.6 [46.9 to 67.9] | 58.0 [48.3 to 67.3]
  rSBA titer >=1.8, Serogroup Y: number analyzed (Participants) | 56 | 66
  rSBA titer >=1.8, Serogroup Y | 62.9 [52.0 to 72.9] | 60.6 [50.7 to 69.8]

3. Secondary Outcome: Group 1: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA and the rSBA and the results were expressed as geometric mean titers.
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and hSBA and rSBA PPAS1 individually consisted of participants for Group 1 visit 1. Only data from the participants analyzed were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
titer
  Day 1: hSBA, Serogroup A | 17.2 [12.6 to 23.3]
  Day 31: hSBA, Serogroup A | 1143 [820 to 1594]
  Day 1: hSBA, Serogroup C | 36.9 [25.7 to 52.9]
  Day 31: hSBA, Serogroup C | 8933 [6252 to 12764]
  Day 1: hSBA, Serogroup Y | 14.6 [10.8 to 19.7]
  Day 31: hSBA, Serogroup Y | 3727 [2908 to 4776]
  Day 1: hSBA, Serogroup W | 29.3 [21.7 to 39.7]
  Day 31: hSBA, Serogroup W | 8656 [6393 to 11721]
  Day 1: rSBA, Serogroup A | 150 [81.7 to 275]
  Day 31: rSBA, Serogroup A | 8454 [6869 to 10405]
  Day 1: rSBA, Serogroup C | 31.5 [18.8 to 52.8]
  Day 31: rSBA, Serogroup C | 20427 [14379 to 29018]
  Day 1: rSBA, Serogroup Y: number analyzed (Participants) | 85
  Day 1: rSBA, Serogroup Y | 64.5 [35.0 to 119]
  Day 31: rSBA, Serogroup Y | 7814 [6111 to 9991]
  Day 1: rSBA, Serogroup W | 49.7 [26.6 to 93.0]
  Day 31: rSBA, Serogroup W | 23354 [17251 to 31615]

4. Secondary Outcome: Group 2: Geometric Mean Titers Against Meningococcal Serogroups A, C, W, and Y
Description: as for outcome 3
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

5. Secondary Outcome: Group 1: Percentage of Participants With hSBA Titer >= 1:4 and >= 1:8
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. hSBA vaccine seroresponse is defined as a post-vaccination titer >= 1:16 for participants with pre-vaccination hSBA titer < 1:8, or a post-vaccination titer >= 4-fold increase at post baseline for participants with pre-vaccination hSBA titer >= 1:8.
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and hSBA PPAS1 consisted of participants for Group 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Day 1: hSBA >=1:4 titer, Serogroup A | 93.2 [85.7 to 97.5]
  Day 31: hSBA >=1:4 titer, Serogroup A | 100 [95.9 to 100]
  Day 1: hSBA >=1:8 titer, Serogroup A | 78.4 [68.4 to 86.5]
  Day 31: hSBA >=1:8 titer, Serogroup A | 98.9 [93.8 to 100]
  Day 1: hSBA >=1:4 titer, Serogroup C | 86.4 [77.4 to 92.8]
  Day 31: hSBA >=1:4 titer, Serogroup C | 97.7 [92.0 to 99.7]
  Day 1: hSBA >=1:8 titer, Serogroup C | 84.1 [74.8 to 91.0]
  Day 31: hSBA >=1:8 titer, Serogroup C | 97.7 [92.0 to 99.7]
  Day 1: hSBA >=1:4 titer, Serogroup Y | 78.4 [68.4 to 86.5]
  Day 31: hSBA >=1:4 titer, Serogroup Y | 100 [95.9 to 100]
  Day 1: hSBA >=1:8 titer, Serogroup Y | 73.9 [63.4 to 82.7]
  Day 31: hSBA >=1:8 titer, Serogroup Y | 100 [95.9 to 100]
  Day 1: hSBA >=1:4 titer, Serogroup W | 95.5 [88.8 to 98.7]
  Day 31: hSBA >=1:4 titer, Serogroup W | 100 [95.9 to 100]
  Day 1: hSBA >=1:8 titer, Serogroup W | 85.2 [76.1 to 91.9]
  Day 31: hSBA >=1:8 titer, Serogroup W | 100 [95.9 to 100]

6. Secondary Outcome: Group 2: Percentage of Participants With hSBA Titer >= 1:4 and >= 1:8
Description: as for outcome 5
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

7. Secondary Outcome: Group 1: Percentage of Participants With rSBA Titer >= 1:8 and >= 1:128
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the rSBA. rSBA vaccine seroresponse is defined as a post-vaccination titer >= 1:32 for participants with pre-vaccination rSBA titer < 1:8, or a post-vaccination titer >= 4-fold increase at post baseline for participants with pre-vaccination rSBA titer >= 1:8.
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and rSBA PPAS1 consisted of participants for Group 1. Only data from the participants analyzed were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Day 1: rSBA >=1:8 titer, Serogroup A | 72.7 [62.2 to 81.7]
  Day 31: rSBA >=1:8 titer, Serogroup A | 100 [95.9 to 100]
  Day 1: rSBA >=1:128 titer, Serogroup A | 64.8 [53.9 to 74.7]
  Day 31: rSBA >=1:128 titer, Serogroup A | 100 [95.9 to 100]
  Day 1: rSBA >=1:8 titer, Serogroup C | 62.5 [51.5 to 72.6]
  Day 31: rSBA >=1:8 titer, Serogroup C | 98.9 [93.8 to 100]
  Day 1: rSBA >=1:128 titer, Serogroup C | 37.5 [27.4 to 48.5]
  Day 31: rSBA >=1:128 titer, Serogroup C | 98.9 [93.8 to 100]
  Day 1: rSBA >=1:8 titer, Serogroup Y: number analyzed (Participants) | 85
  Day 1: rSBA >=1:8 titer, Serogroup Y | 63.5 [52.4 to 73.7]
  Day 31: rSBA >=1:8 titer, Serogroup Y | 98.9 [93.8 to 100]
  Day 1: rSBA >=1:128 titer, Serogroup Y: number analyzed (Participants) | 85
  Day 1: rSBA >=1:128 titer, Serogroup Y | 56.5 [45.3 to 67.2]
  Day 31: rSBA >=1:128 titer, Serogroup Y | 98.9 [93.8 to 100]
  Day 1: rSBA >=1:8 titer, Serogroup W | 58.0 [47.0 to 68.4]
  Day 31: rSBA >=1:8 titer, Serogroup W | 98.9 [93.8 to 100]
  Day 1: rSBA >=1:128 titer, Serogroup W | 50.0 [39.1 to 60.9]
  Day 31: rSBA >=1:128 titer, Serogroup W | 98.9 [93.8 to 100]

8. Secondary Outcome: Group 2: Percentage of Participants With rSBA Titer >= 1:8 and >= 1:128
Description: as for outcome 7
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

9. Secondary Outcome: Group 1: Percentage of Participants With hSBA Titer >=4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and hSBA PPAS1 consisted of participants for Group 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Serogroup A | 93.2 [85.7 to 97.5]
  Serogroup C | 97.7 [92.0 to 99.7]
  Serogroup Y | 98.9 [93.8 to 100]
  Serogroup W | 98.9 [93.8 to 100]

10. Secondary Outcome: Group 2: Percentage of Participants With hSBA Titer >=4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: as for outcome 5
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

11. Secondary Outcome: Group 1: Percentage of Participants With rSBA Titer >=4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Serogroup A | 89.8 [81.5 to 95.2]
  Serogroup C | 96.6 [90.4 to 99.3]
  Serogroup Y: number analyzed (Participants) | 85
  Serogroup Y | 91.8 [83.8 to 96.6]
  Serogroup W | 97.7 [92.0 to 99.7]

12. Secondary Outcome: Group 2: Percentage of Participants With rSBA Titer >=4-Fold Rise From Pre-Vaccination to Post-Vaccination
Description: as for outcome 7
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

13. Secondary Outcome: Group 1: Percentage of Participants With >=0.01 International Units (IU)/mL and >=0.1 IU/mL Anti-Tetanus Antibody Concentration
Description: Anti-tetanus antibodies were measured by diphtheria, tetanus, pertussis multiplexed electrochemiluminescent (DTP-ECL) assay, a multiplexed serological assay that allowed for the simultaneous quantification of human antibodies to 6 specific antigens including diphtheria toxoid, tetanus toxoid, and 4 pertussis antigens: pertussis toxin, filamentous hemagglutinin, fimbriae and pertactin. The captured antibodies were then detected using a sulfotag-conjugated anti-human immunoglobulin (Ig)G conjugate.
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and hSBA PPAS1 consisted of participants for Group 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
percentage of participants
  Day 1: >= 0.01 IU/mL | 100 [95.9 to 100]
  Day 31: >= 0.01 IU/mL | 100 [95.9 to 100]
  Day 1: >= 0.1 IU/mL | 95.5 [88.8 to 98.7]
  Day 31: >= 0.1 IU/mL | 100 [95.9 to 100]

14. Secondary Outcome: Group 2: Percentage of Participants With >=0.01 International Units (IU)/mL and >=0.1 IU/mL Anti-Tetanus Antibody Concentration
Description: as for outcome 13
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

15. Secondary Outcome: Group 1: Geometric Mean Concentrations of Anti-Tetanus Antibody Concentration
Description: Anti-tetanus antibodies were measured by DTP-ECL assay, a multiplexed serological assay that allowed for the simultaneous quantification of human antibodies to 6 specific antigens including diphtheria toxoid, tetanus toxoid, and 4 pertussis antigens: pertussis toxin, filamentous haemagglutinin, fimbriae and pertactin. The captured antibodies were then detected using a sulfotag-conjugated anti-human Ig G conjugate.
Time Frame: Baseline (Day 1) and Day 31 after the administration of a 5-year booster dose
Population: The PPAS is a subset of the FAS and hSBA PPAS1 consisted of participants for Group 1.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 88
IU/mL
  Day 1 | 2.41 [1.77 to 3.30]
  Day 31 | 13.7 [12.0 to 15.7]

16. Secondary Outcome: Group 2: Geometric Mean Concentrations of Anti-Tetanus Antibody Concentration
Description: as for outcome 15
Time Frame: From Baseline (Day 1) until end of the study (approximately 5.5 years)
Reporting Status: Not Posted, anticipated posting 2028-12

17. Secondary Outcome: Group 1: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions (i.e.pre-listed in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination).
Time Frame: Within 30 minutes after vaccination
Population: The Safety analysis set 1 (SafAS 1) consisted of participants who had received the study vaccine 5 years after priming vaccination (Visit 1) and had any safety data available (Group 1).
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 93
Participants | 0

18. Secondary Outcome: Group 1: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions
Description: All noxious and unintended responses to a study vaccine related to any dose was considered adverse reactions (AR). A solicited reaction is an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB. An injection/administration site reaction is an AR at and around the injection/administration site. Injection/administration site reactions are commonly inflammatory reactions. They were considered to be related to the study vaccine administered. Systemic reactions were all ARs that were not injection or administration site reactions and included systemic manifestations such as headache, fever, as well as localized or topical manifestations that are not associated with the vaccination or administration site.
Time Frame: 7 days after vaccination
Population: The SafAS 1 consisted of participants who had received the study vaccine 5 years after priming vaccination (Visit 1) and had any safety data available (Group 1).
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 92
Participants
  Solicited injection site reactions | 67
  Solicited systemic reactions | 45

19. Secondary Outcome: Group 1: Number of Participants With Unsolicited AEs
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE is an observed AE that does not fulfill the conditions of solicited reactions (i.e. pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination). Unsolicited AEs included both serious and non-serious unsolicited AEs.
Time Frame: Within 30 days after vaccination
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 93
Participants | 28

20. Secondary Outcome: Group 1: Number of Participants With Serious AEs (SAEs) and Adverse Event of Special Interest (AESI)
Description: A SAEs is defined as any untoward medical occurrence, at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or other important medical event. An AESI (serious or non-serious) is defined as one of scientific and medical concern specific to the Sponsor's study vaccination or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate.
Time Frame: From the first study vaccine administration up to primary completion date of 09 March 2023, approximately 28 weeks
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | MenACYW: Group 1
Number analyzed (Participants) | 93
Participants
  SAE | 3
  AESI | 0

ADVERSE EVENTS:
Time Frame: From the first study vaccine administration up to primary completion date of 09 March 2023, approximately 28 weeks.
Description: Analysis was performed on SafAS1 population. For 'MenACYW: Group 2', no safety data will be collected as no vaccine administration.
Arm/Group | MenACYW: Group 1 | MenACYW: Group 2
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/93 | 0/0
Other Adverse Events (participants affected / at risk) | 72/93 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW: Group 1 (N=93) | MenACYW: Group 2 (N=0)
Gastroenteritis (Infections and infestations) | 1 (1) | NA
Giardiasis (Infections and infestations) | 1 (1) | NA
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACYW: Group 1 (N=93) | MenACYW: Group 2 (N=0)
Injection Site Erythema (General disorders) | 36 (36) | NA
Injection Site Pain (General disorders) | 60 (60) | NA
Injection Site Swelling (General disorders) | 28 (28) | NA
Malaise (General disorders) | 23 (23) | NA
Pyrexia (General disorders) | 14 (14) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 31 (31) | NA
Headache (Nervous system disorders) | 20 (20) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT04936685/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT04936685/SAP_003.pdf